CLINICAL TRIAL: NCT03452020
Title: Evaluation of the Tyto Thermometer When Used in Clinical Care Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tyto Care Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 790-00038
Record Dates: First submitted 2018-02-14; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Body Temperature Measurement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tyto Thermometer, SoC Thermometer, Predicate IR Th (Other): All the study participants undergo temperature measurements with:
  1. Tyto Thermometer
  2. Standard of Care thermometer
  3. Predicate IR thermometer
  Interventions: Device: Temperature measurementsusing the Tyto thermometer, the standard of care thermometer and the predicate thermometer

INTERVENTIONS:
Device: Temperature measurementsusing the Tyto thermometer, the standard of care thermometer and the predicate thermometer — Temperature measurements using the Tyto thermometer, the standard of care thermometer and the predicate thermometer

SUMMARY:
Patients who present to the Emergency Department will be evaluated for eligibility to the study. Those meeting all the inclusion criteria and none of the exclusion criteria will undergo an informed consent process and will sign a written consent. Within each age group both afebrile and febrile patients will be represented.

The patients will be divided into 3 study groups by age:

Group 1: up to 1 year Group 2: 1 to 5 years Group 3: older than 5 years

The following temperature measurements will be taken:

1. Three temperature measurements using the Tyto thermometer
2. Temperature measurement using the standard of care
3. Three temperature measurements using the predicate device

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, of any age
2. Subject or Parent/Guardian: able to communicate with study personnel;
3. Subject or Parent/Guardian: able to understand the nature of the study and provide written informed consent
4. Subject or Parent/Guardian willing to comply with study procedures

Exclusion Criteria:

1. Cognitive impairment, history of dementia, psychiatric disorders, mental disorders or PDD.
2. Subject or legal guardian unwilling to sign informed consent form
3. Those with signs or recent history of inflammation or infection of the forehead or at the Reference Clinical Test site (site of temperature measurement in any one of the devices used).
4. Subjects currently using cooling blankets, ice on their forehead or fans.
5. Subjects receiving treatment with antipyretics, barbiturates, antipsychotics for the past 3 hours.
6. Subjects receiving current systemic treatment with thyroid preparations, corticosteroids or underwent immunizations during the past 7 days.
7. Subjects with documented illicit drug use or alcoholic intoxication
8. Those participating in a clinical trial of an investigational medicinal product
9. Carriers of multi drug resistant bacteria
10. Pregnancy
11. CTAS score of 1-2

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-06-24 (Estimated); Study Completion 2018-06-24 (Estimated)

PRIMARY OUTCOMES:
Body temperature measurement | a period of no more than 12 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yehezkel Waisman, Prof., Principal Investigator — Director, Department of Emergency Medicine, Schneider Children's Medical Center of Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No